CLINICAL TRIAL: NCT00583622
Title: Bevacizumab Combined With High-Dose Gemcitabine, Docetaxel, Melphalan, and Carboplatin in Patients With Advanced Epithelial Ovarian Cancer
Brief Title: Bevacizumab Plus Gemcitabine, Docetaxel, Melphalan, and Carboplatin in Ovarian Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0368
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-04

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Epithelial Ovarian Cancer; Bevacizumab; Carboplatin; Gemcitabine; Docetaxel; Melphalan
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Bevacizumab; Carboplatin; Docetaxel; Gemcitabine; Melphalan; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + High-Dose Chemotherapy (Experimental): Bevacizumab 5 mg/kg by vein (IV) daily over 90 minutes for 2 Days + Carboplatin 333 mg/m^2 by vein over 2 hours for 3 Days + Docetaxel 300 mg/m^2 by vein over 2 hours for 1 Day + Gemcitabine 1,800 mg/m2 by vein over 3 hours for 4 Days + Melphalan 50 mg/m^2 by vein over 15 minutes for 3 Days + Stem Cell Transplant
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Docetaxel; Drug: Gemcitabine; Drug: Melphalan; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg by vein daily over 90 minutes for 2 Days
  Other Names: Avastin™; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Drug: Carboplatin — 333 mg/m^2 by vein over 2 hours for 3 Days
  Other Names: Paraplatin®
Drug: Docetaxel — 300 mg/m^2 by vein over 2 hours for 1 Day
  Other Names: Taxotere
Drug: Gemcitabine — 1,800 mg/m2 by vein over 3 hours for 4 Days
  Other Names: Gemzar®; Gemcitabine Hyrdrochloride
Drug: Melphalan — 50 mg/m^2 by vein over 15 minutes for 3 Days
Procedure: Stem Cell Transplant — * Stem Cell Removal via apheresis through a central venous catheter (CVC), usually in chest
  * Stem Cell Replacement through CVC over about 30-60 minutes, Day 7 of treatment, following study drug regimen
  Other Names: SCT

SUMMARY:
The goal of this clinical research study is to learn if bevacizumab, when given in combination with gemcitabine, docetaxel, melphalan and carboplatin, or with topotecan, cyclophosphamide and melphalan (if you are older than 60 or have an allergy to carboplatin), can help to control ovarian cancer during a stem cell transplant. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

Carboplatin is designed to damage the DNA (the genetic material) of cancer cells, which may cause them to die.

Melphalan is designed to damage the DNA of cells, which may cause cancer cells to die.

Docetaxel is designed to stop the growth of cancer cells, which may cause the cells to die.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die. It may also help docetaxel, carboplatin, and melphalan to be more effective by stopping tumor cells from repairing damage caused by these drugs.

Topotecan is designed to damage the DNA of cells, which may cause cancer cells to die.

Cyclophosphamide is designed to damage the DNA of cells, which may cause cancer cells to die.

Stem Cell Removal:

Before you begin receiving the study drugs, you will have apheresis done to collect some of your stem cells as a part of your standard of care. Apheresis is the process of removing part of the blood (such as platelets or white blood cells) from the body in order to remove certain elements, such as stem cells. Then, the rest of the blood is returned back to your body.

Apheresis will be done through a central venous catheter (CVC), usually in the chest. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain these procedures to you in more detail, and you will be required to sign a separate consent form for each procedure.

Your stem cells will be put back in your body after you finish receiving gemcitabine, docetaxel, melphalan, and carboplatin.

To prevent clotting, citrate (a blood thinner) will be added to the CVC during the apheresis procedure.

Study Drug Administration:

If you are found to be eligible to take part in this study, 2 weeks before your admission to the hospital (about 3 weeks before the stem cell transplant), you will receive bevacizumab through a the CVC over 45 minutes.

On Day 1 of your stay in the hospital, you will receive bevacizumab through the CVC over 45 minutes.

As part of standard mouth care, you will be asked to do mouthwashes 4 times a day (for 2 minutes each time) with caphosol (artificial saliva) followed by glutamine. Fifteen (15) minutes after each caphosol mouthwash, you will swish glutamine around in your mouth and gargle for 2 minutes, then spit it out. Do not swallow it.

On Day 2, through the CVC, you will receive gemcitabine over 3 hours and docetaxel over 2 hours. If you are allergic to carboplatin or older than 60 you will receive topotecan over 30 minutes.

On Day 3-5, through the CVC, you will receive gemcitabine over 3 hours, melphalan over 15 minutes, and carboplatin over 2 hours.

On Day 6, you will not receive any study drugs.

On Day 7, you will receive the stem cells through the CVC over about 30-60 minutes.

Starting the day after your stem cell transplant, as part of standard care, you will receive granulocyte-colony stimulating factor (G-CSF or filgrastim) as an injection under your skin daily, starting 1 day after the transplant, until your blood cell levels return to normal.

Starting 2 days after your transplant until 10 days after your transplant, you will receive methylprednisolone 2 times a day.

If you are allergic to carboplatin or older than 60:

On Day 1 of your stay in the hospital, you will receive bevacizumab through the CVC over 45 minutes.

On Day 2-4, through the CVC, you will receive cyclophosphamide over 2 hours and topotecan over 30 minutes. Each time you receive cyclophosphamide, you will also receive mesna to decrease the risk of bleeding in the bladder.

On Day 5-6, through the CVC, you will receive melphalan over 30 minutes and topotecan over 30 minutes.

On Day 7, you will not receive any study drugs.

On Day 8, you will receive the stem cells through the CVC over about 30-60 minutes.

Starting the day after your stem cell transplant, as part of standard care, you will receive G-CSF (filgrastim) as an injection under your skin daily, starting 1 day after the transplant, until your blood cell levels return to normal.

Study Visits:

At least once a week after the transplant, and then about 30, 60, and 100 days after your stem cell transplant, the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam.
* You will be checked for possible reactions to the treatment, including graft-versus-host disease (GVHD) and graft failure. Graft failure occurs when donor cells may not be able to grow and multiply in your body. If this happens, there will be a high risk of infections and/or bleeding.
* Blood (about 3 tablespoons) will be drawn for routine tests and to check for tumor markers to check the status of the disease.
* Urine will be collected for routine tests.
* You will have a pelvic exam, if your doctor thinks it is needed.
* You will have an ECHO, if your doctor thinks it is needed.
* You will have a lung function test, if your doctor thinks it is needed.
* You will have CT scans of your chest, abdomen, and pelvis to check the status of the disease, if your doctor thinks it is needed.
* You will have a positron emission tomography - computed tomography (PET-CT) scan to check the status of the disease. A PET-CT is CT scan taken after a small amount of radioactive glucose (sugar) is injected into a vein to find cancer cells in the body.

These tests and procedures may be performed more often, if your doctor thinks it is needed.

End-of-Treatment Visit:

About 6 and 12 months after your stem cell transplant, then once a year after that (if your doctor thinks it is needed), the study visit tests and procedures listed above will be repeated.

Length of Study:

You will be off study after about 6 months. You will be taken off study early if the disease gets worse, if not enough stem cells can be collected, or if you experience any intolerable side effects.

Long-Term Follow-up:

If your doctor thinks it is necessary, you may have follow-up visits.

This is an investigational study. Bevacizumab is FDA approved and commercially available for the treatment of colorectal cancer. Gemcitabine, docetaxel, melphalan, and carboplatin are all FDA-approved and commercially available for the treatment of ovarian cancer. The use of bevacizumab with gemcitabine, docetaxel, melphalan, and carboplatin is investigational.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - <70.
2. Patients with advanced ovarian, fallopian or primary peritoneal cancer in second or later complete remission, or untreated or refractory relapse, defined as relapse within 6 months of prior platinum treatment or lack of response to salvage treatment.
3. No evidence of small bowel obstruction, as determined by CT scan of the abdomen and pelvis with oral and rectal contrast, within 30 days before the initiation of study treatment.
4. Adequate renal glomerular and tubular function, as defined by estimated serum creatinine clearance >=60 ml/min, and urinary protein excretion <=500 mg/day.
5. Adequate hepatic function, as defined by serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) <=3 * upper limit of normal (ULN); serum bilirubin and alkaline phosphatase <=2 * ULN or considered not clinically significant.
6. Adequate pulmonary function with Forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and Carbon Monoxide Diffusing Capacity (DLCO) >=50% of predicted, corrected for volume or hemoglobin.
7. Adequate cardiac function with left ventricular ejection fraction >=45%. No uncontrolled arrhythmias or symptomatic cardiac disease.
8. Zubrod performance status <2.

Exclusion Criteria:

1. Failure to collect more than 3 * 10e6 CD34+ stem cells/kg body weight
2. Patients with unresolved grade 3 or greater non-hematologic toxicity from previous therapy. Patients with grade 2 toxicity will be eligible at the discretion of the principal investigator.
3. Major surgery within 30 days before the initiation of study treatment
4. Radiotherapy within 21 days prior to initiation of study treatment
5. Patients with active Central Nervous System (CNS) disease.
6. Evidence of acute or chronic active hepatitis or cirrhosis. If positive hepatitis serology, discuss with Principal Investigator and consider liver biopsy.
7. Uncontrolled infection, including HIV or HTLV-1 infection.
8. Aspirin (> 325 mg/day) use within 10 days before initiation of study treatment.
9. Ongoing uncontrolled hypertension (>140/90 mm Hg on medication).
10. Non-healing wound or significant traumatic injury within 30 days before the initiation of study treatment
11. Previous autologous or allogeneic stem cell transplant during the past year.
12. Positive Beta HCG test in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yago Nieto, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 19, 2007 to January 11, 2012. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: One participant of the 13 enrolled did not receive treatment and was excluded from the study.
Period: Overall Study
Arm/Group | Bevacizumab + High-Dose Chemotherapy
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab + High-Dose Chemotherapy
Number analyzed (Participants) | 12
Age Continuous [Median (Full Range); unit: years] | 47 [33 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Event-Free (EF) Rate
Description: Percent of participants free of relapse or disease progression at end of 6 months. Event-free survival estimated from the first day of High-dose chemotherapy (day-6) until tumor progression, relapse, or death from any cause.
Time Frame: Up to 6 Months
Population: Due to the small number of patients treated, 12 out of 30 planned, an analysis was not possible.
Arm/Group | Bevacizumab + High-Dose Chemotherapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Participant Response
Description: Number of participants evaluated using Response to Treatment in Solid Tumors (RECIST) with definitions of Complete Response (CR): disappearance of all target lesions; and, Partial Response: at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Maintained Continued CR: participants who entered study in a CR and maintained CR post study treatment. Evaluations once a week till Day +30, then Days 30, 60, and 100 then at 6 months or until disease progression.
Time Frame: Up to 6 months
Population: One participant was not evaluable for response as participant expired prior to performing restaging evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + High-Dose Chemotherapy
Number analyzed (Participants) | 12
percentage of participants
  Complete Response (CR) | 33.3
  Maintained Continued CR | 42.0
  Partial Response (PR) | 8.3
  No Response | 8.3
  Not Evaluable | 8.3

ADVERSE EVENTS:
Time Frame: 3 years and six months
Arm/Group | Bevacizumab + High-Dose Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + High-Dose Chemotherapy (N=12)
Death (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab + High-Dose Chemotherapy (N=12)
Mucositis (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 9 (9)
Elevated Bilirubin (Hepatobiliary disorders) | 2 (2)
Enterococcus Infection (Infections and infestations) | 2 (2)
Neutropenic Fever (Infections and infestations) | 9 (9)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Skin Rash (Skin and subcutaneous tissue disorders) | 8 (8)
Fever (General disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No